CLINICAL TRIAL: NCT00073008
Title: A Phase 2 Multicenter Trial Comparing Two Schedules of GW572016 as First or Second Line Monotherapy in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer With Either Bronchioloalveolar Carcinoma or No Smoking History
Brief Title: A Study Of Oral GW572016 In Advanced Or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment was stopped due to lack of efficacy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF20014; NCT00084955 (obsolete NCT alias)
Record Dates: First submitted 2003-11-13; First posted 2003-11-17 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: EGFR; ErbB1; ErbB2; metastatic; lapatinib; Her-2/neu; protein kinase inhibitor; BAC; GW572016; Advanced; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lapatinib (Other): Randomized, open-label, parallel group, 2-stage study to evaluate and compare 2 dose schedules (1500 mg once daily and 500 mg twice daily) of oral lapatinib.
  Interventions: Drug: GW572016 (lapatinib)

INTERVENTIONS:
Drug: GW572016 (lapatinib) — tyrosine kinase inhibitor

SUMMARY:
This study was designed to evaluate and compare the efficacy of two dose schedules of an oral investigational drug for the treatment of advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Subjects must have histologically confirmed advanced (incurable stage IIIB or IV according to the International Staging System, [Mountain, 1997] Non-Small Cell Lung Cancer (NSCLC) at primary diagnosis or relapsed after curative-intent surgery. Only patients with either (1) the histological subtypes of adenocarcinoma with BAC (Bronchioloalveolar) features or pure BAC (as defined by the 1999 World Health Organization criteria) or, (2) never smokers (i.e. smoked <100 cigarettes in lifetime) with any histology of NSCLC (squamous, adenocarcinoma, lifetime) with any histology of NSCLC (squamous, adenocarcinoma,
* Patients can have had a maximum of 1 prior systemic therapy (chemotherapy or biologic therapy) for NSCLC that ended at least 3 weeks prior to enrollment. Patients that have had adjuvant cytotoxic chemotherapy that ended at least 3 months prior to enrollment are eligible. Prior surgery and radiotherapy are permitted. Patients should recover from acute side effects of radiation before enrollment (3-4 weeks). Concurrent radiotherapy is prohibited;
* Archived tumor tissue available for evaluation of genetic and intra-tumoral protein or mRNA expression levels of relevant biomarkers. A minimum of 10 slides of archived tumor tissue is required; however, 15 slides should be sent, if available. For patients diagnosed on the basis of pleural effusions, efforts should be made to provide as many slides as possible made with cells obtained from pleural aspirates. Results of biomarkers will not be used to determine subject eligibility for the study;
* Measurable lesion(s) according to RECIST (e.g., ≥15 mm with conventional techniques (medical photograph [skin or oral lesion], palpation, plain X-ray, CT, MRI, or ≥10 mm with spiral CT scan);
* At least 1 measurable lesion located outside of the prior radiation field or, if located within the prior field of irradiation, is increasing in size;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1;
* Life expectancy of ≥ 12 weeks;
* ≥ 18 years old;
* A female is eligible to enter and participate in this study if she is of: • Non-childbearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation, women who had a hysterectomy, women who are post-menopausal, or women who have had both ovaries surgically removed); or • Childbearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhea (even severe), women who are perimenopausal, and young women who have begun to menstruate. Women of childbearing potential must have a negative serum pregnancy test at screening, and agree to 1 of the following: a Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of GW572016 until 28 days after the final dose of GW572016; or b Consistent and correct use of 1 of the following acceptable methods of birth control: 1. Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; or 2. Implants of levonorgestrel 3. Injectable progestogen 4. Any intrauterine device (IUD) with a documented failure rate of less than 1% per year; or 5. Oral contraceptives (either combined or Progestogen only) 6. Barrier methods including diaphragm or condom with a spermicide
* Able to swallow and retain oral medication;
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram. Subjects with known history of uncontrolled or symptomatic echocardiogram. Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure are not eligible;
* Have adequate organ function as defined in Table 1 Baseline Laboratory Values for Inclusion;
* Subjects must complete all screening assessments as outlined in the protocol.

Exclusion Criteria:

* Malabsorption Syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible;
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety;
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug;
* Active or uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* Uncontrolled angina, arrhythmias, or congestive heart failure. Patients whose symptoms are under control are eligible.
* Known history of or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or antiseizure medication for ≥ 3 months prior to study enrollment. Routine screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases;
* Concurrent cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, and tumor embolization).
* Concurrent treatment with an investigational agent or participation in another clinical trial
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of GW572016;
* Prior therapy with any ErbB1 and/or ErbB2 inhibitor;
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GW572016.
* Has taken/received the following inhibitors of CYP3A4 within the specified number of days prior to the first dose of study medication: Seven (7) days: antibiotics (clarithromycin, erythromycin, troleandomycin), antiretrovirals (delavirdine), protease inhibitors (ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir), systemic antifungals (itraconazole, ketoconazole, voriconazole, fluconazole (doses of 200 mg/day and above)), antidepressants (nefazodone, fluovoxamine), calcium channel blockers (verapamil, diltiazem), gastrointestinal (cimetidine, aprepitant), and grapefruit or its juice. Six (6) months: amiodarone.
* Has taken/received the following inducers of CYP3A4 within fourteen (14) days prior to the first dose of study medication: glucocorticoids (dexamethasone or dexamethasone equivalent dose > 1.5mg/day (see chart in Section 7.2 for conversion), anticonvulsants (phenytoin, carbamazepine, phenobarbital), efavirenz, nevirapine, antibiotics (rifampin (rifampicin), rifabutin, rifapentine), St. John's Wort and modafinil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2003-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (23):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Gainsville, Florida
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Houma, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Nyack, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Houston, Texas
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Lévis, Quebec

REFERENCES:
- [Background] Colin F Spraggs, Laura R Parham, Christine M. Hunt and Colin T Dollery. Characterisation of lapatinib-associated DILI cases by Class II HLA and UGT1A1*28 genotypes. [Clin Pharmacol Ther]. 2012;
- [Background] Ross HJ, Blumenschein GR Jr, Aisner J, Damjanov N, Dowlati A, Garst J, Rigas JR, Smylie M, Hassani H, Allen KE, Leopold L, Zaks TZ, Shepherd FA. Randomized phase II multicenter trial of two schedules of lapatinib as first- or second-line monotherapy in patients with advanced or metastatic non-small cell lung cancer. Clin Cancer Res. 2010 Mar 15;16(6):1938-49. doi: 10.1158/1078-0432.CCR-08-3328. Epub 2010 Mar 9. PMID 20215545

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib 1500 mg QD: Oral lapatinib 1500 mg once daily (QD)
- Lapatinib 500 mg BID: Oral lapatinib 500 mg twice daily (BID)
Period: Overall Study
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Started | 65 | 66
Completed | 3 | 3
Not Completed | 62 | 63
Not completed — Missing | 6 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 46 | 47
Not completed — "Other" selected on Case Report Form | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.03) | 65.2 (10.56) | 65.1 (11.27)
Gender [Count of Participants; unit: Participants]
  Female | 33 | 40 | 73
  Male | 32 | 26 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54 | 56 | 110
  Black | 4 | 1 | 5
  Asian | 4 | 5 | 9
  American Hispanic | 2 | 4 | 6
  Other | 1 | 0 | 1
Histology at diagnosis [Number; unit: Participants] — Type of lung cancer
  Participants
    Squamous cell | 9 | 3 | 12
    Bronchioloalveolar carcinoma (BAC) | 3 | 2 | 5
    Adenocarcinoma with BAC features | 8 | 13 | 21
    Adenocarcinoma without BAC features | 34 | 43 | 77
    Other non-small cell lung cancer type | 5 | 1 | 6
    Other | 4 | 2 | 6
    Missing | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response in the Targeted Population Through the End of Treatment
Description: Disease progression and tumor response (number of participants achieving a complete response [CR] or partial response [PR]), using standardized criteria (Response evaluation criteria in solid tumors). CR, disappearance of all target lesions; PR, 30% decrease in the sum of the longest diameter of target lesions; progressive disease, 20% increase in the sum of the longest diameter of target lesions; stable disease, small changes that do not meet above criteria. Disease assessment was done at baseline and then every 8 weeks after starting treatment, until the participant discontinued treatment.
Time Frame: Baseline and then every 8 weeks through end of treatment
Population: Targeted Population: all randomized participants who received at least one dose of study drug and had either the histological subtypes of adenocarcinoma with bronchioloalveolar carcinoma features or pure bronchioloalveolar carcinoma, or were never smokers with any histology of non-small cell lung cancer (NSCLC)
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 24 | 32
participants
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 5 | 9
  Progressive disease | 18 | 20
  Missing | 1 | 3

2. Other Pre Specified Outcome: Tumor Response in the Non-Targeted Population Through the End of Treatment
Description: Baseline and then every 8 weeks through end of treatment (end of treatment for each participant was dependent on when the participant withdrew from study therapy due to disease progression, an adverse event or participant decision)
Time Frame: Baseline and then every 8 weeks through end of treatment
Population: Non-Targeted Population: all randomized participants who received at least one dose of study drug but who did not meet the criteria for inclusion in the Targeted Population.
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 41 | 34
participants
  Complete response | 0 | 0
  Partial response | 1 | 0
  Stable disease | 10 | 6
  Progressive disease | 27 | 25
  Missing | 3 | 3

3. Secondary Outcome: Progression-free Survival (PFS) at Four Months in the Targeted Population
Description: Percentage of participants in the Targeted Population, at 4 months after starting study drug, who were alive and without disease progression.
Time Frame: From randomization and then every 8 weeks up to four months
Population: Targeted Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 24 | 32
percentage of participants | 34.5 | 19.7
Statistical Analysis 1: Comparison: Lapatinib 1500 mg QD; Test type: Superiority or Other; Kaplan-Meier estimate = 34.5, 95% CI [13.7 to 55.4] — Percentage of surviving participants who were progression free 4 months after the date of randomization
Statistical Analysis 2: Comparison: Lapatinib 500 mg BID; Test type: Superiority or Other; Kaplan-Meier estimate = 19.7, 95% CI [2.9 to 36.4] — Percentage of surviving participants who were progression free 4 months after the date of randomization

4. Secondary Outcome: Progression-free Survival (PFS) at Four Months in the Non-Targeted Population
Description: Percentage of participants in the Non-Targeted Population, at 4 months after starting study drug, who were alive and without disease progression.
Time Frame: From randomization and then every 8 weeks up to four months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 41 | 34
percentage of participants | 27.1 | 18.3
Statistical Analysis 1: Comparison: Lapatinib 1500 mg QD; Test type: Superiority or Other; Kaplan-Meier estimate = 27.1, 95% CI [11.9 to 42.3] — Percentage of surviving participants who were progression free 4 months after the date of randomization
Statistical Analysis 2: Comparison: Lapatinib 500 mg BID; Test type: Superiority or Other; Kaplan-Meier estimate = 18.3, 95% CI [3.9 to 32.6] — Percentage of surviving participants who were progression free 4 months after the date of randomization

5. Secondary Outcome: The Number of Participants Who Showed Certain Biomarkers in Their Serum or Tumor Tissue
Description: To further characterize the participant population, these biomarkers could be tested: serum levels of ErbB1 and ErbB2; intra-tumoral expression of ErbB1, ErbB2, etc.; mutations in ErbB1, ErbB2, and k-ras. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, serum biomarkers were not analyzed.
Time Frame: From randomization to disease progression (for serum biomarkers) or until analyses of tumor tissue samples
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacokinetics (PK) of Lapatinib
Description: To characterize the PK (absorption, distribution, metabolism, and excretion) of the study drug lapatinib in the participant population. PK is defined as the concentration of drug in a participant's blood at certain time points after the drug was taken by mouth. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, pharmacokinetics were not analyzed.
Time Frame: From randomization to time of PK period completed: Day 1 (first dose) and Days 2, 28, and 29 while participant was on study drug
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacogenetics (PgX)
Description: To (1) investigate the relationship between genetic variants in specific genes and the absorption, distribution, metabolism, and excretion (pharmacokinetics) of lapatinib, and to (2) investigate the relationship between genetic variants in select genes in DNA and the response (safety, efficacy, and tolerability) to lapatinib. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, pharmacogenetics were not analyzed.
Time Frame: From randomization at every 4-week assessment through end of treatment
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Quality of Life
Description: Standard survey forms were completed by the participant at scheduled assessments to find out how the participant felt while on study. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, quality of life was not analyzed.
Time Frame: Baseline and then every 4 weeks through end of treatment
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Response
Description: Time from randomization until first documented evidence of partial or complete tumor response, measured using standard criteria (RECIST). Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, time to response was not analyzed.
Time Frame: From randomization and then every 8 weeks to time of response to study drug
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Duration of Response
Description: For those participants who show a complete or partial response, duration of response would be time from first documented evidence of response (complete or partial response by RECIST) until disease progression or death, if sooner. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, duration of response was not analyzed.
Time Frame: Time from first documented evidence of response to study treatment and then every 8 weeks until disease progression or death
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Tumor Progression
Description: Time from randomization until the first documented sign of disease progression or death due to any cause, if sooner. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, time to tumor progression was not analyzed.
Time Frame: From randomization and then every 8 weeks to disease progression or death
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Overall Survival
Description: Overall survival is measured as the time from randomization until death due to any cause. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, overall survival was not analyzed.
Time Frame: From randomization and then every 8 weeks while on study drug and then every 3 months as follow-up until death
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Review of Non-small Cell Lung Cancer (NSCLC) Histology (Cell Type) Using an Independent Review
Description: Comparison of the specific cell type (histology) of non-small cell lung cancer from participant's tissue samples, as determined by local pathologist, to the type determined by an independent pathologist. Based on the interim analysis at the end of Stage 1, and predefined stopping rules for futility, further enrollment into the study was stopped due to lack of efficacy on both treatment arms; therefore, NSCLC histology was not analyzed.
Time Frame: Anytime from Baseline through end of study
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Lapatinib 1500 mg QD | Lapatinib 500 mg BID
Serious Adverse Events (participants affected / at risk) | 15/65 | 17/66
Other Adverse Events (participants affected / at risk) | 64/65 | 63/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg QD (N=65) | Lapatinib 500 mg BID (N=66)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Cardiac disorders) | 2 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea hemorrhagic (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg QD (N=65) | Lapatinib 500 mg BID (N=66)
Diarrhea (Gastrointestinal disorders) | 39 | 33
Rash (Skin and subcutaneous tissue disorders) | 31 | 27
Fatigue (General disorders) | 24 | 20
Nausea (Gastrointestinal disorders) | 25 | 16
Anorexia (Metabolism and nutrition disorders) | 17 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 12
Constipation (Gastrointestinal disorders) | 10 | 11
Vomiting (Gastrointestinal disorders) | 15 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 10
Dysgeusia (Nervous system disorders) | 7 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Dizziness (Nervous system disorders) | 6 | 7
Pyrexia (General disorders) | 9 | 4
abdominal pain (Gastrointestinal disorders) | 6 | 6
insomnia (Psychiatric disorders) | 9 | 3
pruritus (Skin and subcutaneous tissue disorders) | 5 | 7
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 5
edema peripheral (General disorders) | 5 | 5
chest pain (General disorders) | 4 | 5
headache (Nervous system disorders) | 6 | 3
weight decreased (Investigations) | 7 | 2
alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
asthenia (General disorders) | 4 | 4
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 4
flatulence (Gastrointestinal disorders) | 3 | 5
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
anaemia (Blood and lymphatic system disorders) | 4 | 3
anxiety (Psychiatric disorders) | 5 | 2
chills (General disorders) | 5 | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
nasopharyangitis (Infections and infestations) | 3 | 4
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 5
upper respiratory tract infection (Infections and infestations) | 3 | 4
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
chest discomfort (General disorders) | 2 | 4
dyspepsia (Gastrointestinal disorders) | 1 | 5
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
neuropathy peripheral (Nervous system disorders) | 4 | 2
pneumonia (Infections and infestations) | 2 | 4
stomatitis (Gastrointestinal disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
Based on interim analysis and predefined stopping rules for futility, the study was discontinued due to lack of efficacy. At that time, no additional participants were added; enrolled participants could continue on treatment, following the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.